CLINICAL TRIAL: NCT01943292
Title: A Phase I Dose Escalation Study to Evaluate the Safety and Pharmacokinetics of VS-6063, a Focal Adhesion Kinase Inhibitor, in Japanese Subjects With Non-Hematologic Malignancies
Brief Title: Phase I Dose Escalation Study of VS-6063 in Japanese Subjects With Non-Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-6063-102
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2016-01

CONDITIONS: Non Hematologic Cancers
Keywords: Focal Adhesion Kinase inhibitor; FAK inhibitor; Cancer Stem Cells; CSC
MeSH Terms: interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Defactinib (Experimental): Oral defactinib (VS-6063) administered twice a day (BID) during a 21 day cycle.
  Interventions: Drug: Defactinib

INTERVENTIONS:
Drug: Defactinib
  Other Names: VS-6063

SUMMARY:
This is a phase I, open-label, dose-escalation trial of defactinib (VS-6063), a focal adhesion kinase inhibitor, in Japanese patients with non-hematologic malignancies. The purpose of this study is to assess the safety (including the recommended phase 2 dose), the pharmacokinetics, and the anti-cancer activity of defactinib (VS-6063).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed and dated informed consent prior to initiation of any study procedures.
* Age ≥ 20 years.
* Subject must be of Japanese descent.
* Subjects must have a histopathologically confirmed diagnosis of a non-hematologic malignancy.
* Subjects must have no further standard of care options or have refused standard therapy.
* All persistent clinically significant toxicities from prior chemotherapy must be ≤ Grade 1.
* ECOG performance status of 0 or 1, measured within 72 hours before the start of treatment.
* Predicted life expectancy of ≥ 3 months.
* Adequate renal function [creatinine ≤ 1.5x ULN (upper limit of normal)] or GFR of ≥ 50mL/min.
* Adequate hepatic function (total bilirubin ≤ 1.5x ULN for the institution; AST [aspartate transaminase] and ALT [alanine transaminase] ≤ 3x ULN, or ≤ 5x ULN if due to liver involvement by tumor).
* Adequate bone marrow function (hemoglobin ≥ 9.0 g/dL; platelets ≥ 100 x109 cells/L; absolute neutrophil count ≥ 1.5x109 cells/L).
* Corrected QT interval (QTc) < 470 ms (as calculated by the Fridericia correction formula).
* Negative pregnancy test for women of child-bearing potential. (A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant except for women who have undergone permanent contraceptive surgery or are postmenopausal (defined as the absence of menstruation for at least 12 months without other medical reasons).
* Men and women of child bearing potential must agree to use adequate birth control throughout their participation in the study and for 90 days following the last study treatment.
* Willing and able to participate in the trial and comply with all trial requirements.

Exclusion Criteria:

* Gastrointestinal (GI) condition which could interfere with the swallowing or absorption of study medication.
* Uncontrolled or severe concurrent medical condition (including uncontrolled brain metastases). Stable brain metastases either treated or being treated with a stable dose of steroids/ anticonvulsants, with no dose change within 28 days prior to the first dose of study drug, will be allowed.
* History of upper gastrointestinal bleeding, ulceration, or perforation within 12 months prior to the first dose of study drug.
* Known history of stroke or cerebrovascular accident within 6 months prior to the first dose of study drug.
* Subjects with known infection with human immunodeficiency virus (HIV) or Acquired Immune Deficiency Syndrome (AIDS) (testing not required).
* Subjects with known Hepatitis B or C (Including known seropositivity Hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV antibody).
* Subjects being actively treated for a secondary malignancy.
* Cancer-directed therapy (chemotherapy, radiotherapy, hormonal therapy, biologic or immunotherapy, etc.) within 28 days of the first dose of study drug or 5 half-lives, whichever is shorter.
* Major surgery within 28 days prior to the first dose of study drug.
* Use of an investigational drug within 28 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug. A minimum of 10 days between termination of the investigational drug and administration of the study treatment is required. In addition, any drug-related toxicity except alopecia should have recovered to grade 1 or less.
* Women who are pregnant or breastfeeding.
* Any evidence of serious active infections.
* Uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months prior to study treatment, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, or cardiac amyloidosis.
* Known history of malignant hypertension
* Uncontrolled intercurrent illness including symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2014-06-09 (Actual); Study Completion 2014-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, m, Study Chair — Verastem, Inc.
Locations (1):
- Kinki University Hospital, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 02Sep2013; Last subject enrolled 07Jan2014; all patients enrolled at one site in Japan.
Pre-assignment Details: There were no significant events and approaches for overall study. There was one screen failure.
Groups:
- Defactinib 200 mg Bid: 200 mg bid (twice a day) po (by mouth) defactinib
- Defactinib 400 mg Bid: 400 mg bid po defactinib
- Defactinib 600 mg Bid: 600 mg bid po defactinib
Period: Overall Study
Arm/Group | Defactinib 200 mg Bid | Defactinib 400 mg Bid | Defactinib 600 mg Bid
Started | 3 | 3 | 3
Completed Cycle 1 | 3 | 3 | 3
Completed Treatment | 3 | 3 | 3
Completed Follow-Up | 2 | 3 | 3
Completed | 2 | 3 | 3
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Defactinib 200 mg Bid: 200 mg po bid defactinib
- Defactinib 400 mg Bid: 400 mg po bid defactinib
- Defactinib 600 mg Bid: 600 mg po bid defactinib
- Total: Total of all reporting groups
Arm/Group | Defactinib 200 mg Bid | Defactinib 400 mg Bid | Defactinib 600 mg Bid | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (6.51) | 67.0 (7.21) | 53.7 (16.56) | 60.4 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2
  Male | 3 | 3 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Assess the Safety and Tolerability of Defactinib (VS-6063) in Japanese Subjects With Non-hematologic Malignancies
Description: A composite by dose level to include incidence of AEs, SAEs, dose interruptions and dose reductions as a measure of safety and tolerability. Abnormal Clinical significant laboratory results, ECG measurements, vital signs measurement, physical examination findings, and ECOG performance status were captured as adverse events.
  The severity of AEs were evaluated according to CTCAE (Common Toxicity Criteria for Adverse Effects) 4.03
Time Frame: From start of treatment to end of treatment, an expected average of 12 weeks
Measure: Number; unit: participants
Arm/Group | Defactinib 200 mg Bid | Defactinib 400 mg Bid | Defactinib 600 mg Bid
Number analyzed (Participants) | 3 | 3 | 3
participants
  At least 1 TEAE (treatment emergent AE) | 3 | 3 | 3
  At least 1 TEAE related to study drug | 3 | 3 | 3
  Non-Lab TEAE with Severity ≥ Grade 3 | 0 | 0 | 0
  Lab TEAE with Severity ≥ Grade 3 | 1 | 0 | 0
  At least 1 Serious TEAE | 0 | 0 | 0
  Dose Interruptions | 1 | 1 | 0
  Dose Reductions | 0 | 0 | 0

2. Secondary Outcome: Define the Maximum Tolerated Dose (MTD), if Achieved, and Establish the Recommended Phase 2 Dose (RP2D) of Defactinib (VS-6063) in Japanese Subjects.
Description: The RP2D will be determined based on the MTD of defactinib (VS-6063) as determined by number of participants with dose limiting toxicities (DLTs) related to defactinib.
Time Frame: From start of treatment to end of cycle 1 (21 day cycles)
Measure: Number; unit: mg
Arm/Group | Defactinib 200 mg Bid | Defactinib 400 mg Bid | Defactinib 600 mg Bid
Number analyzed (Participants) | 3 | 3 | 3
mg | NA — There were no DLTs. MTD was not reached. RP2D is 400 mg bid. | NA — There were no DLTs. MTD was not reached. RP2D is 400 mg bid. | NA — There were no DLTs. MTD was not reached. RP2D is 400 mg bid.

3. Secondary Outcome: Assess the Pharmacokinetics, Metabolism and Elimination of Defactinib (VS-6063) in Plasma and Urine.
Description: PK parameters, including but not limited to plasma concentration, AUC (Area Under Curve) 0-t, Cmax, Tmax, and T1/2. Total 24-hour urine output will be collected in conjunction with PK sampling to assess the elimination of defactinib (VS-6063) and its potential metabolites.
Time Frame: Time points at Day 1 and Day 15 in Cycle 1
Reporting Status: Not Posted

4. Secondary Outcome: Evaluate the Efficacy (Response Rate and Progression-free Survival) of Subjects Treated With Defactinib (VS-6063).
Description: Response rate and progression-free survival, as determined by Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1
Time Frame: Every 8 weeks up to end of treatment, an expected average of 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) include all events (related and unrelated) from the time patient doses through 30 days post last dose of study treatment
Description: The systematic method was through regular investigator assessment and regular laboratory testing.
Arm/Group | Defactinib 200 mg Bid | Defactinib 400 mg Bid | Defactinib 600 mg Bid
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Defactinib 200 mg Bid (N=3) | Defactinib 400 mg Bid (N=3) | Defactinib 600 mg Bid (N=3)
Blood Bilirubin Increased (Investigations) | 3 | 2 | 2
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 2 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 3
Headache (Nervous system disorders) | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 1 | 0
Blood Phosphorus Increased (Investigations) | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
There were no limitations of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site is not able to publish any clinical trial results without first seeking permission from Verastem.